CLINICAL TRIAL: NCT05239728
Title: A Multicenter, Double-blind, Randomized Phase 3 Study to Compare the Efficacy and Safety of Belzutifan (MK-6482) Plus Pembrolizumab (MK-3475) Versus Placebo Plus Pembrolizumab in the Adjuvant Treatment of Clear Cell Renal Cell Carcinoma (ccRCC) Post Nephrectomy (MK-6482-022)
Brief Title: A Study of Belzutifan (MK-6482) Plus Pembrolizumab (MK-3475) Versus Placebo Plus Pembrolizumab in Participants With Clear Cell Renal Cell Carcinoma Post Nephrectomy (MK-6482-022)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6482-022; MK-6482-022 (Other: MSD); LITESPARK-022 (Other: MSD); jRCT2051220030 (Registry Identifier: jRCT); 2023-505023-31-00 (Registry Identifier: EU CT); U1111-1290-7346 (Registry Identifier: UTN); 2021-003436-92 (EudraCT Number)
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Renal Cell
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1(PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2); Hypoxia inducible factor 2 alpha (HIF-2 alpha); Hypoxia inducible factor 2α (HIF-2α)
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — belzutifan; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan + Pembrolizumab (Experimental): Participants receive belzutifan 120 mg orally once daily (QD) for up to approximately 54 weeks PLUS pembrolizumab 400 mg via intravenous (IV) infusion once every 6 weeks (Q6W) for up to 9 administrations (up to approximately 54 weeks).
  Interventions: Drug: Belzutifan; Biological: Pembrolizumab
- Placebo + Pembrolizumab (Experimental): Participants receive placebo orally QD for up to approximately 54 weeks PLUS pembrolizumab 400 mg via IV infusion once Q6W for up to 9 administrations (up to approximately 54 weeks).
  Interventions: Biological: Pembrolizumab; Drug: Placebo

INTERVENTIONS:
Drug: Belzutifan — Three 40 mg tablets given as a single oral 120 mg dose.
  Other Names: MK-6482; PT2977; WELIREG™
  Arms: Belzutifan + Pembrolizumab
Biological: Pembrolizumab — 400 mg via IV infusion
  Other Names: MK-3475; Keytruda®
Drug: Placebo — Oral tablet
  Arms: Placebo + Pembrolizumab

SUMMARY:
The purpose of this study is to assess the efficacy and safety of oral belzutifan (MK-6482) plus intravenous (IV) pembrolizumab (MK-3475) compared to placebo plus pembrolizumab, in the adjuvant treatment of Clear Cell Renal Cell Carcinoma (ccRCC) post nephrectomy.

The primary study hypothesis is that belzutifan plus pembrolizumab is superior to placebo plus pembrolizumab with respect to disease-free survival (DFS).

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of RCC with clear cell component per American Joint Committee on Cancer (AJCC) (8th Edition), with or without sarcomatoid features
* Has intermediate-high risk, high risk, or M1 no evidence of disease (NED) RCC as defined by the following pathological tumor-node metastasis and tumor grading:

  1. Intermediate-high risk RCC: pT2, Grade 4 or sarcomatoid, N0, M0; pT3, any grade, N0, M0
  2. High risk RCC: pT4, any Grade N0, M0; pT any stage, any Grade, N+, M0
  3. M1 NED RCC participants who present not only with the primary kidney tumor but also solid, isolated, soft tissue metastases that can be completely resected at one of the following: the time of nephrectomy (synchronous) or, ≤2 years from nephrectomy (metachronous)
* Has undergone complete resection of the primary tumor (partial or radical nephrectomy) and complete resection of solid, isolated, soft tissue metastatic lesion(s) in M1 NED participants
* Must have undergone a nephrectomy and/or metastasectomy ≤12 weeks prior to randomization
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 within 10 days before randomization.
* Male participants must agree to continue contraception at least 7 days after the last dose of belzutifan/placebo
* Female participants of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of pembrolizumab or at least 30 days after last dose of belzutifan/placebo, whichever occurs last
* Has adequate organ function

Exclusion Criteria:

* Has had a major surgery, other than nephrectomy plus resection of preexisting metastases for M1 NED participants, within 4 weeks prior to randomization
* Has a pulse oximeter reading <92% at rest, requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
* Has clinically significant cardiovascular disease within 6 months from first dose of study intervention
* Has other clinically significant disorders such as: serious active nonhealing wound/ulcer/bone fracture; requirement for hemodialysis or peritoneal dialysis
* Has preexisting brain or bone metastatic lesions
* Has received prior systemic therapy for RCC
* Has received prior radiotherapy for RCC
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention; administration of killed vaccines are allowed
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has a known additional malignancy (other than RCC treated with nephrectomy and/or metastasectomy) that is progressing or has required active treatment within the past 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs); replacement therapy is allowed
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection, requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection, a known history of Hepatitis B or known active Hepatitis C virus infection
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-10-28 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | Up to approximately 54 months
  DFS is defined as the time from randomization to the first documented local recurrence, or occurrence of distant kidney cancer metastasis(es) as assessed by investigator, or death due to any cause, whichever occurs first. The DFS for all participants will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 89 months
  OS is defined as the time from randomization to death due to any cause.
Number of Participants Who Experience at Least One Adverse Event (AE) | Up to approximately 66 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 54 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued the study due to an AE will be reported.
Disease Recurrence-Specific Survival 1 (DRSS1) | Up to approximately 54 months
  DRSS1 is defined as the time from randomization to the first documented local recurrence of RCC as assessed by the investigator. For DRSS1, only local recurrence is counted as an event.
Disease Recurrence-Specific Survival 2 (DRSS2) | Up to approximately 54 months
  DRSS2 is defined as the time from randomization to the first documented local recurrence with visceral lesion or occurrence of distant kidney cancer metastasis(es) with visceral lesion, whichever occurs first, as assessed by investigator.
Change From Baseline in Health-Related Quality-of-Life (HRQoL) Using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Items 29 and 30 Score | Baseline (Day 1) and up to approximately 36 months
  The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of participants with cancer. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. The change from baseline in EORTC QLQ-C30 Items 29 and 30 combined scores will be presented.
Change From Baseline in Physical Functioning Using the EORTC QLQ-C30 Items 1- 5 Score | Baseline (Day 1) and up to approximately 36 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher scores indicate a worse level of function. Change from baseline in the score of EORTC QLQ-C30 Items 1-5 will be presented.
Change From Baseline in Role Functioning Using the EORTC QLQ-C30 Items 6 and 7 Score | Baseline (Day 1) and up to approximately 36 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to questions about their role functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Higher score indicate a worse level of function. Change from baseline in the score of EORTC QLQ-C30 Items 6-7 will be presented.
Change From Baseline in Disease Symptoms Using the Functional Assessment of Cancer Therapy-Kidney Symptom Index-Disease-related Symptoms (FKSI-DRS) Items 1-9 Score | Baseline (Day 1) and up to approximately 36 months
  The FKSI-DRS index consists of a 9-item questionnaire that assesses the extent of participant symptoms from kidney cancer. Responses are scored on a 5-point scale (0=Not at all to 4=Very much) and summed to generate an index symptom score. These scores can range from 0 to 36, with a higher score indicating more favorable kidney cancer symptom status. Change from baseline in the score of FKSI-DRS Items 1-9 will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (285):
- United States (37):
  - Mayo Clinic in Arizona - Phoenix ( Site 3554), Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center ( Site 3567), Duarte, California
  - Moores Cancer Center-Clinical Trials Office- Genitourinary ( Site 3516), La Jolla, California
  - UCLA Hematology/Oncology - Westwood (Building 200 Suite 140)-Department of Urology/Institute of Uro ( Site 3520), Los Angeles, California
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 3518), Orange, California
  - Stanford Cancer Center ( Site 3523), Palo Alto, California
  - University of Colorado Anschutz Medical Campus ( Site 3514), Aurora, Colorado
  - Intermountain Health St. Mary's Regional Hospital ( Site 3562), Grand Junction, Colorado
  - Georgetown University Medical Center ( Site 3534), Washington D.C., District of Columbia
  - University of Miami Hospital and Clinics, Sylvester Cancer Center-Cancer Research Services ( Site 3517), Miami, Florida
  - Moffitt Cancer Center ( Site 3540), Tampa, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital-Research ( Site 3515), Marietta, Georgia
  - Parkview Research Center at Parkview Regional Medical Center ( Site 3526), Fort Wayne, Indiana
  - Johns Hopkins Hospital-Sidney Kimmel Comprehensive Cancer Center- GU Oncology ( Site 3549), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 3571), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center-Cancer Clinical Trials Office ( Site 3572), Boston, Massachusetts
  - Dana-Farber Cancer Institute-GU ( Site 3505), Boston, Massachusetts
  - Cancer and Hematology Centers of Western Michigan ( Site 3502), Grand Rapids, Michigan
  - Washington University-Internal Medicine/Oncology ( Site 3531), St Louis, Missouri
  - St. Vincent Frontier Cancer Center-Research ( Site 3506), Billings, Montana
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists ( Site 3550), Omaha, Nebraska
  - Englewood Hospital and Medical Center ( Site 3557), Englewood, New Jersey
  - Rutgers Cancer Institute of New Jersey ( Site 3541), New Brunswick, New Jersey
  - Monter Cancer Center ( Site 3560), Lake Success, New York
  - Icahn School of Medicine at Mount Sinai ( Site 3539), New York, New York
  - Memorial Sloan Kettering Cancer Center ( Site 3568), New York, New York
  - University of Rochester Medical Center ( Site 3528), Rochester, New York
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive C ( Site 3507), Columbus, Ohio
  - MidLantic urology ( Site 3501), Bala-Cynwyd, Pennsylvania
  - Fox Chase Cancer Center-GU Oncology ( Site 3535), Philadelphia, Pennsylvania
  - Sanford Cancer Center ( Site 3551), Sioux Falls, South Dakota
  - The West Clinic, PLLC dba West Cancer Center ( Site 3522), Germantown, Tennessee
  - Urology Associates ( Site 3512), Nashville, Tennessee
  - UT Southwestern Medical Center ( Site 3529), Dallas, Texas
  - University of Texas MD Anderson Cancer Center-Urology ( Site 3569), Houston, Texas
  - Inova Schar Cancer Institute ( Site 3525), Fairfax, Virginia
  - Seattle Cancer Care Alliance-Renal/Melanoma/MCC ( Site 3524), Seattle, Washington
- Australia (7):
  - Blacktown Hospital ( Site 0002), Blacktown, New South Wales
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 0003), Macquarie University, New South Wales
  - Tamworth Hospital-North West Cancer Centre ( Site 0006), North Tamworth, New South Wales
  - Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Site 0001), Brisbane, Queensland
  - Lyell McEwin Hospital-Oncology Clinical Trials Unit ( Site 0008), Elizabeth Vale, South Australia
  - Austin Health-Cancer Clinical Trials Centre ( Site 0005), Heidelberg, Victoria
  - Fiona Stanley Hospital-Medical Oncology ( Site 0004), Murdoch, Western Australia
- Brazil (7):
  - Hospital São Carlos-Oncocentro Ce ( Site 0104), Fortaleza, Ceará
  - Centro Avançado de Tratamento Oncológico- CENANTRON-Clinical Research ( Site 0105), Belo Horizonte, Minas Gerais
  - Instituto do Câncer e Transplante de Curitiba ( Site 0102), Curitiba, Paraná
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0103), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0101), Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Ribeirão Preto ( Site 0112), Ribeirão Preto, São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo ( Site 0111), São Paulo
- Bulgaria (3):
  - MBAL Uni Hospital-Department of Medical Oncology ( Site 0204), Panagyurishte, Pazardzhik
  - MHAT Serdika-Second Department of Medical Oncology ( Site 0203), Sofia, Sofia (stolitsa)
  - Complex Cancer Center Plovdiv-First Medical Oncology Department ( Site 0205), Plovdiv
- Canada (8):
  - Arthur J.E. Child Comprehensive Cancer Centre ( Site 3706), Calgary, Alberta
  - BC Cancer Vancouver-Clinical Trials Unit ( Site 3707), Vancouver, British Columbia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 3710), Hamilton, Ontario
  - Victoria Hospital & Children's Hospital - London Health Scie-London Regional Cancer Program ( Site 3705), London, Ontario
  - Princess Margaret Cancer Centre ( Site 3703), Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 3708), Montreal, Quebec
  - McGill University Health Centre ( Site 3709), Montreal, Quebec
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 3701), Québec, Quebec
- Chile (8):
  - Clínica Puerto Montt ( Site 0309), Port Montt, Los Lagos Region
  - Oncocentro Valdivia ( Site 0312), Valdivia, Los Ríos Region
  - FALP-UIDO ( Site 0302), Santiago, Region M. de Santiago
  - Oncovida ( Site 0306), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0305), Santiago, Region M. de Santiago
  - James Lind Centro de Investigacion del Cancer ( Site 0307), Temuco, Región de la Araucanía
  - ONCOCENTRO APYS-ACEREY ( Site 0301), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 0303), Antofagasta
- China (30):
  - Afflilated Hospital of Bengbu Medical College-Urology Surgery ( Site 0438), Bengbu, Anhui
  - Second Affiliated hospital of Anhui Medical University-Urology ( Site 0416), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science-Urinary Surgery ( Site 0435), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Urinary Surgery ( Site 0406), Beijing, Beijing Municipality
  - First Medical Center of Chinese PLA General Hospital ( Site 0415), Beijing, Beijing Municipality
  - Peking University First Hospital-Urology ( Site 0407), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 0414), Chongqing, Chongqing Municipality
  - Army Medical Center of People's Liberation Army ( Site 0439), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University-Urology ( Site 0445), Fuzhou, Fujian
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 0403), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-Urology Surgery ( Site 0402), Guangzhou, Guangdong
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE-Urology Surgery ( Site 0417), Guangzhou, Guangdong
  - Henan Cancer Hospital-Urology ( Site 0441), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology-oncology ( Site 0423), Wuhan, Hubei
  - Wuhan Union Hospital ( Site 0430), Wuhan, Hubei
  - Hubei Cancer Hospital-Urinary surgery ( Site 0419), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 0421), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( Site 0424), Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University ( Site 0443), Nanchang, Jiangxi
  - The First affiliated hospital of Nanchang University (Xianghu campus) ( Site 0432), Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 0431), Xi'an, Shaanxi
  - Fudan University Shanghai Cancer Center-Urology department ( Site 0401), Shanghai, Shanghai Municipality
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 0418), Shanghai, Shanghai Municipality
  - Huadong Hospital Affiliated to Fudan University ( Site 0405), Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University-Urology Surgery ( Site 0410), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 0422), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 0428), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital-Urology ( Site 0426), Hangzhou, Zhejiang
  - Ningbo First Hospital-Urology ( Site 0433), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Urology Surgery ( Site 0425), Wenzhou, Zhejiang
- Colombia (4):
  - Clinica de la Costa S.A.S. ( Site 0506), Barranquilla, Atlántico
  - Administradora Country S.A. - Clinica del Country ( Site 0504), Bogotá, Bogota D.C.
  - Sociedad De Oncologia Y Hematologia Del Cesar-Oncology ( Site 0505), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0501), Montería, Departamento de Córdoba
- Czechia (7):
  - Fakultni Nemocnice u sv. Anny v Brne-Onkologicko-chirurgicke oddeleni ( Site 0603), Brno, Brno-mesto
  - Masarykuv onkologicky ustav-Klinika komplexni onkologicke pece ( Site 0605), Brno, Brno-mesto
  - Fakultni nemocnice Ostrava-Klinika onkologicka ( Site 0606), Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 0601), Olomouc, Olomoucký kraj
  - Fakultni Thomayerova nemocnice-Onkologicka klinika 1. LF UK ( Site 0602), Prague, Praha 4
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 0607), Prague, Praha 5
  - Fakultni nemocnice Hradec Kralove-Klinika onkologie a radioterapie ( Site 0604), Hradec Králové
- Finland (5):
  - Oulun yliopistollinen sairaala ( Site 0802), Oulu, North Ostrobothnia
  - Kuopion Yliopistollinen Sairaala-Syöpäkeskus ( Site 0804), Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala ( Site 0805), Tampere, Pirkanmaa
  - Turku University Hospital ( Site 0801), Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus) ( Site 0803), Helsinki, Uusimaa
- France (9):
  - Institut de cancérologie Strasbourg Europe (ICANS) ( Site 0903), Strasbourg, Alsace
  - CENTRE LEON BERARD-Medical oncology ( Site 0902), Lyon, Auvergne-Rhône-Alpes
  - ROC37 ( Site 0910), Chambray-lès-Tours, Centre-Val de Loire
  - CHU Besançon-Medical oncology ( Site 0904), Besançon, Doubs
  - Centre Hospitalier Universitaire de Rennes - Hôpital Pontchaillou ( Site 0908), Rennes, Ille-et-Vilaine
  - Centre Hospitalier Universitaire d'Angers-Urology ( Site 0901), Angers, Maine-et-Loire
  - Hôpital Saint-Louis ( Site 0905), Paris
  - Hôpital Européen Georges Pompidou-Service d'Oncologie Médicale ( Site 0906), Paris
  - Gustave Roussy ( Site 0907), Villejuif, Île-de-France Region
- Germany (16):
  - Hegau-Bodensee-Klinikum Singen ( Site 1016), Singen, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen ( Site 1002), Tübingen, Baden-Wurttemberg
  - klinikum rechts der isar der technischen universität münchen-Urologische Klinik und Poliklinik ( Site 1003), Munich, Bavaria
  - Universitätsklinikum Aachen ( Site 1024), Aachen, North Rhine-Westphalia
  - Universitätsklinikum Bonn ( Site 1006), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf ( Site 1017), Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 1004), Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus ( Site 1005), Münster, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes-Klinik fuer Urologie und Kinderurologies ( Site 1020), Homburg, Saarland
  - Universitaetsklinikum Carl Gustav Carus Dresden-Klinik und Poliklinik für Urologie ( Site 1021), Dresden, Saxony
  - Krankenhaus Martha-Maria Halle-Dölau-Klinik für Urologie, Kinderurologie und urologische Onkologie ( Site 1008), Halle, Saxony-Anhalt
  - SRH Wald-Klinikum Gera ( Site 1015), Gera, Thuringia
  - Universitätsklinikum Jena ( Site 1007), Jena, Thuringia
  - Charité Universitaetsmedizin Berlin - Campus Mitte ( Site 1022), Berlin
  - Helios Klinikum Berlin-Buch ( Site 1011), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf-Onkologisches Zentrum ( Site 1001), Hamburg
- Greece (5):
  - Alexandra Hospital-ONCOLOGY DEPT. ( Site 1102), Athens, Attica
  - Metropolitan Hospital-2nd Oncology Dept ( Site 1104), Athens, Attica
  - ATTIKON GENERAL UNIVERSITY HOSPITAL ( Site 1101), Chaïdári, Attica
  - Euromedica General Clinic Thessaloniki-Oncology Unit ( Site 1103), Thessaloniki
  - European Interbalkan Medical Center-Oncology Department ( Site 1105), Thessaloniki
- Hungary (5):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ ( Site 1319), Szeged, Csongrád megye
  - Petz Aladar Egyetemi Oktato Korhaz-Onkológiai Osztály ( Site 1321), Győr, Győr-Moson-Sopron
  - Országos Onkológiai Intézet-Urogenitális Tumorok és Klinikai Farmakológiai Osztály ( Site 1316), Budapest, Pest County
  - Somogy Megyei Kaposi Mór Oktató Kórház-Oncology center ( Site 1311), Kaposvár, Somogy County
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 1310), Debrecen
- Ireland (4):
  - St. Vincent's University Hospital ( Site 1401), Dublin, Dublin
  - Tallaght University Hospital ( Site 1402), Dublin, Dublin
  - Cork University Hospital ( Site 1404), Cork
  - Beaumont Hospital, Dublin-Cancer Clinical Trials & Research Unit ( Site 1403), Dublin
- Israel (6):
  - Soroka Medical Center ( Site 1505), Beersheba
  - Rambam Health Care Campus-Oncology ( Site 1502), Haifa
  - Hadassah Medical Center-Oncology ( Site 1506), Jerusalem
  - Rabin Medical Center-Oncology ( Site 1503), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 1504), Ramat Gan
  - Sourasky Medical Center-Oncology ( Site 1501), Tel Aviv
- Italy (10):
  - A.O.U.C. Policlinico di Bari ( Site 1607), Bari, Apulia
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori-Oncologia Medica ( Site 1603), Meldola, Emilia-Romagna
  - Fondazione Policlinico Universitario Agostino Gemelli-Medical Oncology ( Site 1604), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1608), Milan, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga-SCDU Oncologia Medica ( Site 1602), Orbassano, Piedmont
  - Azienda Ospedaliera Universitaria Careggi-SOD ONCOLOGIA MEDICA ( Site 1601), Florence, Tuscany
  - Azienda USL 8 di Arezzo-Medical Oncology ( Site 1610), Arezzo
  - IRCCS - AOU di Bologna-Oncologia Medica Ardizzoni ( Site 1605), Bologna
  - Ospedale San Raffaele-Oncologia Medica ( Site 1606), Milan
  - Azienda Ospedaliera Santa Maria Terni-SC Oncologia ( Site 1609), Terni
- Japan (21):
  - Fujita Health University Hospital ( Site 1709), Toyoake, Aichi-ken
  - National Cancer Center Hospital East ( Site 1704), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 1718), Sakura, Chiba
  - Ehime University Hospital ( Site 1714), Tōon, Ehime
  - Sapporo Medical University Hospital ( Site 1702), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 1701), Sapporo, Hokkaido
  - Kanagawa Cancer Center ( Site 1703), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 1712), Kashihara, Nara
  - Bell Land General Hospital ( Site 1710), Sakai, Osaka
  - The University of Osaka Hospital ( Site 1711), Suita, Osaka
  - Hamamatsu University Hospital ( Site 1708), Hamamatsu, Shizuoka
  - Toranomon Hospital ( Site 1706), Minato-ku, Tokyo
  - Toyama University Hospital ( Site 1713), Toyoma, Toyama
  - Kyushu University Hospital ( Site 1715), Fukuoka
  - Kagoshima University Hospital ( Site 1719), Kagoshima
  - Kumamoto University Hospital ( Site 1716), Kumamoto
  - Okayama University Hospital ( Site 1720), Okayama
  - Nippon Medical School Hospital ( Site 1705), Tokyo
  - Tokyo Women's Medical University Adachi Medical Center ( Site 1717), Tokyo
  - Keio University Hospital ( Site 1707), Tokyo
  - Wakayama Medical University Hospital ( Site 1721), Wakayama
- Malaysia (3):
  - University Malaya Medical Centre ( Site 1804), Lembah Pantai, Kuala Lumpur
  - Hospital Pulau Pinang ( Site 1806), George Town, Pulau Pinang
  - Sarawak General Hospital-Radiotherapy Unit ( Site 1805), Kuching, Sarawak
- Mexico (12):
  - Terapias Integrales del Riñon SA de CV ( Site 1910), Guadalajara, Jalisco
  - Hospital Civil Fray Antonio Alcalde-Oncology ( Site 1906), Guadalajara, Jalisco
  - BRCR Global Mexico - Guadalajara-Research ( Site 1908), Guadalajara, Jalisco
  - INSTITUTO NACIONAL DE CANCEROLOGIA ( Site 1902), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran-Oncologia y Hematologia ( Site 1912), Mexico City, Mexico City
  - Filios Alta Medicina ( Site 1903), Monterrey, Nuevo León
  - iCan Oncology Center Centro Medico AVE ( Site 1901), Monterrey, Nuevo León
  - Hospital H+ Queretaro-Cuidados Oncológicos ( Site 1905), Querétaro City, Querétaro
  - BRCR Global Mexico - Queretaro-SMIQ ( Site 1907), Querétaro City, Querétaro
  - Centro de Oncología Personalizada ( Site 1911), Culiacán, Sinaloa
  - Centro de Investigacion Clinica de Oaxaca ( Site 1904), Oaxaca City
  - Oncocenter ( Site 1909), Puebla City
- Netherlands (15):
  - Ziekenhuis Rijnstate-Rijnstate Centrum Oncologisch Onderzoek ( Site 3113), Arnhem, Gelderland
  - Radboudumc ( Site 3120), Nijmegen, Gelderland
  - Maastricht UMC+ ( Site 3104), Maastricht, Limburg
  - Amphia Ziekenhuis, locatie Breda Molengracht ( Site 3103), Breda, North Brabant
  - Maxima Medisch Centrum, locatie Eindhoven ( Site 3116), Eindhoven, North Brabant
  - Amsterdam UMC, locatie AMC ( Site 3105), Amsterdam, North Holland
  - Tergooiziekenhuizen, locatie Hilversum ( Site 3102), Hilversum, North Holland
  - Spaarne Gasthuis - Hoofddorp-Oncology ( Site 3107), Hoofddorp, North Holland
  - Isala, locatie Zwolle-Oncology ( Site 3111), Zwolle, Overijssel
  - Haaglanden MC - locatie Antoniushove ( Site 3117), Leidschendam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Vlietland ( Site 3101), Schiedam, South Holland
  - Haga Ziekenhuis locatie Leyweg-Oncology ( Site 3108), The Hague, South Holland
  - University Medical Center Groningen ( Site 3121), Groningen
  - St. Antonius Ziekenhuis, locatie Utrecht-Interne geneeskunde ( Site 3112), Utrecht
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 3106), Utrecht
- Auckland City Hospital ( Site 2003), Auckland, New Zealand
- Poland (12):
  - Przychodnia Lekarska KOMED ( Site 2304), Konin, Greater Poland Voivodeship
  - Szpital Kliniczny im. Przemienienia Panskiego Uniwersytetu M-chemotherapy department ( Site 2312), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2307), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MICS Centrum Medyczne Torun ( Site 2305), Torun, Kuyavian-Pomeranian Voivodeship
  - Szpital Wojewódzki im. Świętego Lukasza SP ZOZ w Tarnowie ( Site 2311), Tarnów, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 2313), Siedlce, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 2303), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 2301), Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu ( Site 2306), Przemyśl, Podkarpackie Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu ( Site 2309), Wrocław, Silesian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie-Oddzial Dzienny Chemioterapii ( Site 2302), Koszalin, West Pomeranian Voivodeship
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne ( Site 2315), Szczecin, West Pomeranian Voivodeship
- Romania (6):
  - Cardiomed SRL Cluj-Napoca ( Site 2406), Cluj-Napoca, Cluj
  - Amethyst Radiotherapy Center-Oncologie Medicala ( Site 2405), Florești, Cluj
  - Centrul de Oncologie Sfantul Nectarie-Medical ( Site 2401), Craiova, Dolj
  - Radiology Therapeutic Center-Oncology ( Site 2404), Otopeni, Ilfov
  - Cabinet Medical Oncomed ( Site 2403), Timișoara, Timiș County
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L ( Site 2407), Bucharest
- Singapore (2):
  - National Cancer Centre Singapore ( Site 3601), Singapore, Central Singapore
  - National University Hospital ( Site 3602), Singapore, South West
- South Korea (4):
  - National Cancer Center-Center for Urologic Cancer ( Site 2604), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital-Urology ( Site 2602), Seongnam, Kyonggi-do
  - Asan Medical Center-Oncology ( Site 2601), Songpagu, Seoul
  - Samsung Medical Center ( Site 2603), Seoul
- Spain (8):
  - Institut Català d'Oncologia (ICO) - Girona ( Site 2707), Girona, Gerona
  - Hospital Universitario Ramón y Cajal-Medical Oncology ( Site 2710), Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre-Medical Oncology ( Site 2708), Madrid, Madrid, Comunidad de
  - Fundación Instituto Valenciano de Oncología ( Site 2705), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Departamento de Oncologia- VHIO ( Site 2702), Barcelona
  - Hospital Lucus Augusti-Oncology ( Site 2706), Lugo
  - Hospital Clinico San Carlos-Oncology Department ( Site 2703), Madrid
  - Hospital Universitario Virgen de la Victoria-Phase II-III-IV Trials ( Site 2709), Málaga
- Sweden (3):
  - Karolinska Universitetssjukhuset Solna ( Site 2802), Stockholm, Stockholm County
  - Akademiska sjukhuset-Blod- och tumörsjukdomar ( Site 2803), Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset ( Site 2801), Gothenburg, Västra Götaland County
- Taiwan (8):
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 2905), Kaohsiung Niao Sung Dist, Kaohsiung
  - Tri-Service General Hospital ( Site 2908), Taipei City, Taipei
  - Kaohsiung Veterans General Hospital ( Site 2901), Kaohsiung City
  - China Medical University Hospital-Department of Urology ( Site 2907), Taichung
  - Taichung Veterans General Hospital ( Site 2902), Taichung
  - National Taiwan University Hospital ( Site 2904), Taipei
  - Taipei Veterans General Hospital ( Site 2903), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Urology ( Site 2906), Taoyuan District
- Thailand (4):
  - Chulalongkorn University ( Site 3005), Bangkok, Bangkok
  - Ramathibodi Hospital ( Site 3001), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 3002), Bangkok, Bangkok
  - Songklanagarind hospital ( Site 3004), Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (8):
  - Istanbul Universitesi Cerrahpasa-Internal Diseases ( Site 3204), Istanbul- Fatih, Istanbul
  - Baskent University Dr. Turgut Noyan Research and Training Center-ONCOLOGY ( Site 3208), Adana
  - Ankara Gülhane Eitim ve Aratrma Hastanesi-Oncology ( Site 3207), Ankara
  - Ankara University Hospital Cebeci ( Site 3209), Ankara
  - Hacettepe Universitesi-oncology hospital ( Site 3203), Ankara
  - Ankara Bilkent Şehir Hastanesi-oncology ( Site 3206), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 3201), Istanbul
  - Ege University Medicine of Faculty-Medical Oncology ( Site 3202), Izmir
- United Kingdom (7):
  - Royal Free Hospital ( Site 3304), London, England
  - The Christie NHS Foundation Trust ( Site 3301), Manchester, England
  - City Hospital, Nottingham University Hospitals ( Site 3303), Nottingham, England
  - Beatson West of Scotland Cancer Centre-Clinical Trials Unit ( Site 3305), Glasgow, Glasgow City
  - Charing Cross Hospital ( Site 3302), London, Hammersmith and Fulham
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 3307), London, London, City of
  - Singleton Hospital ( Site 3306), Swansea

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26232&tenant=MT_MSD_9011